CLINICAL TRIAL: NCT05148195
Title: An Open Label, Multi-cohort, Multicenter Phase II Study to Evaluate the Efficacy and Safety of Envofolimab in Combination With BD0801 Injection With/Without Chemotherapy in Patients With Advanced Solid Tumors
Brief Title: A Phase II Study of Envofolimab and BD0801 With/Without Chemotherapy in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to the sponsor's research and development strategy adjustment.
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B02B00302-KN035-201
Record Dates: First submitted 2021-11-15; First posted 2021-12-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Docetaxel; Irinotecan; Leucovorin; 5-fluorouridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: Solid tumor (Experimental): Envofolimab（300mg，Q3W）+BD0801（2mg/kg，Q3W）
  Interventions: Drug: Envofolimab; Drug: BD0801
- B: HCC (Experimental): Envofolimab（300mg，Q3W）+BD0801（2mg/kg，Q3W）
  Interventions: Drug: Envofolimab; Drug: BD0801
- D：NSCLC (Experimental): Envofolimab（300mg，Q3W）+BD0801（2mg/kg，Q3W）+Docetaxel(75mg/m2，Q3W)
  Interventions: Drug: Envofolimab; Drug: BD0801; Drug: Docetaxel
- D：CRC (Experimental): Envofolimab（200mg，Q2W）+BD0801（2mg/kg，Q2W）+FOLFIRI（Irinotecan 180 mg/m2，Leucovorin 400mg/m2，5-Fluorouridine 2400 mg/m2，Q2W）
  Interventions: Drug: Envofolimab; Drug: Irinotecan; Drug: Leucovorin calcium; Drug: 5-Fluorouridine

INTERVENTIONS:
Drug: Envofolimab — 300mg，Q3W (arm A,B and C)or 200mg, Q2W(arm D)
Drug: BD0801 — 2mg/kg，Q3W(armA, B and C) or 2mg/kg，Q2W
  Arms: A: Solid tumor; B: HCC; D：NSCLC
Drug: Docetaxel — 75mg/m2，Q3W
  Arms: D：NSCLC
Drug: Irinotecan — 180 mg/m2，Q2W
  Arms: D：CRC
Drug: Leucovorin calcium — 400mg/m2，Q2W
  Arms: D：CRC
Drug: 5-Fluorouridine — 2400 mg/m2，Q2W
  Arms: D：CRC

SUMMARY:
This is an open label, multi-cohort, multicenter Phase II study, the purpose of this study is to assess the efficacy and safety of envofolimab in combination with BD0801 injection with/without chemotherapy for the treatment of advanced solid tumors

DETAILED DESCRIPTION:
The efficacy of immune checkpoint inhibitors combined with antivascular agents has been preliminarily demonstrated in a variety of solid tumors. Based on the huge clinical needs, the efficacy of envofolimab combined with BD0801 in patients with advanced hepatocellular carcinoma, non-small cell lung cancer and advanced colorectal cancer deserves further exploration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent;
2. Age≥18 age years old, male or female;
3. Patients diagnosed with unresectable or advanced solid tumors confirmed by histopathology or cytology; Cohort A: Patients must have progressed on standard of therapy, patients with NSCLC, CRC and HCC (include intrahepatic cholangiocarcinoma or mixed hepatocellular carcinoma-cholangiocarcinoma in safety run-in phase) are enrolled preferentially; Cohort B: Patients with histopathologically or cytologically or clinically diagnosed advanced HCC (Barcelona Clinic Liver Cancer (BCLC) Stage C; or BCLC Stage B patients who are not suitable for locoregional therapy (such as TACE) may also be enrolled), Child-Pugh liver function grade A and patients received at least one standard first-line systemic treatment and no more than 3 systemic regimens for HCC; Cohort C: Histologically confirmed NSCLC (except for patients with central and cavernous lung squamous cell carcinoma). Patients received at least one standard first line systemic treatment are required, if patients with EGFR、ALK or ROS1 gene positive, first line of target therapy will be required ( if patients with known EGFR mutation, they should be T790M negative or with osimertinib treatment failure); C1: Required prior anti-PD-1/PD-L1 therapy. C2: Never used prior anti-PD-1/PD-L1 therapy. Cohort D: Patients with advanced CRC confirmed with histology, the results of tissue samples must meet any of the following (1. the test result of immunohistochemistry is mismatch repair protein integrity (pMMR) 2. the test result of NGS is MSI-L or MSS 3 the test of result of PCR is MSI-L or MSS). Has received the oxaliplatin and 5-Fu containing regimen for the treatment of metastatic tumors.
4. ECOG score 0 or 1;
5. At least one measurable lesion as per RECIST V1.1;
6. Normal major organ and marrow functions as defined and no blood transfusion and blood product within 2 weeks before screening, no use of hematopoietic stimulating factors;
7. Life expectancy≥12 weeks;
8. Women of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose. Male or female patients of childbearing potential voluntarily use effective contraceptive methods from signing the informed consent form to 6 months after initiation of the study drug, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. All female patients are considered to be of childbearing potential unless they are postmenopausal (continuous menopause for 12 month), had undergone artificial menopause, or had undergone surgical sterilization (e.g., hysterectomy, surgical adnexectomy);

Exclusion Criteria:

1. Patients who have participated in clinical trials of other investigational drugs or investigational devices within 28 days prior to the first dose or received any systemic treatments within 2 weeks, include but not limited chemotherapy, radiotherapy (palliative radiotherapy is allowed at least 1 week before the study drug treatment), targeted therapy, Chinese herbal medicine or proprietary Chinese medicine for cancer control;
2. Patients with a history of Envofolimab or BD0801 treatment;
3. Patients who have ascites requiring drainage or diuretic treatment or pleural effusion or pericardial effusion requiring drainage and/or accompanied by shortness of breath within 2 weeks before the first dose of study drug treatment;
4. Cholangiocarcinoma, mixed cell carcinoma, or fibroblastic layer cell carcinoma are known for Cohort B;
5. Patients with other active malignancies within 2 years prior to the first administration of the study drug randomization, curable localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical carcinoma in situ, and carcinoma in situ of the breast can be included in the group;
6. Patients whose toxicity and side effects (due to previous anticancer treatments) have not recovered to≤grade 1, unless such AE is not considered to pose safety risks (such as hair loss and neuropathy≤grade 2 caused by oxaliplatin)
7. Patients with previous and current central nervous system (CNS)metastasis;
8. Patients with a history of hepatic encephalopathy;
9. Patients with active tuberculosis (TB), who are receiving anti-TB treatment or received anti-TB treatment within 3 months prior the first study drug administration;
10. Abdominal fistula, gastrointestinal perforation, abdominal abscess and intestinal obstruction with clinical symptoms (including occlusive disease);
11. Receipt of live or attenuated live vaccines 4 weeks prior to the first study drug treatment;
12. Suffer from any disease that requires corticosteroids within 2 weeks prior to the first study drug administration, except for local corticosteroids or dose of prednisone or equivalent drugs≤ 10mg/ day;
13. Patients with previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-associated pneumonia, and severe impairment of lung function that may interfere with the detection and management of suspected drug-related lung toxicity;
14. Patients with known activity or autoimmune diseases or history. Except subjects with vitiligoare not requiring systemic treatment within 2 years prior the first study drug, type 1 diabetes mellitus, hypothyroidism requiring only hormone replacement therapy, pituitaritis and adrenal cortical insufficiency requiring only physiological hormone replacement therapy or psoriasis who do not require systemic treatment may be allowed;
15. Major surgery before enrollment or expected major surgery during the study period;
16. Severe unhealed wound, ulcers or fractures;
17. The current or recent (within 10 days before the first dose of study medication) use of aspirin for 10 days (> 325 mg/day) or other known to inhibit platelet function of NSAIDs; a history bleeding disorders or thrombosis within 6 months before the first study drug administration;
18. Patients with clinically significant cardiovascular diseases；
19. Cardiac function: Left ventricular ejection fraction (LVEF)<50%;
20. Human immunodeficiency virus (HIV) antibodies or acquired immune deficiency syndrome (AIDS);
21. Active hepatitis B (HBsAg positive and HBV- DNA ≥ULN) or hepatitis C (HCV antibody positive and quantitative HCV-RNA≥ULN);
22. Pregnant or lactating women during the study;
23. Patients with a history of allergy to studied drugs or similar drugs or excipients;
24. Other conditions that researchers consider inappropriate for inclusion;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Part I: MTD（Maximum tolerable dose）or RD（Recommended dose） | 6 months
  MTD: A maximum dose of acceptable safety, at least 6 patients treated with this dose, and less than 1/3 of patients experienced DLT(Dose limited toxicity).
  RD:The following will be taken into account to make decision about RD: MTD, if is reached; PK characteristics, efficacy and safety results.
Part II: ORR(Objective Response Rate ) by investigator | 1.5 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
DOR(Duration Of Response) by investigator | 1.5 years
  Measured from the date of partial or complete response to therapy until the disease progression based on RECIST v1.1criteria.
PFS(Progression Free Survival) by investigator | 1.5 years
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigator according to the RECIST1.1 criteria
DCR(Disease Control Rate) by investigator | 1.5 years
  Proportion of subjects who have a complete or partial response, or stable disease relative to baseline as assessed by investigator according to RECIST 1.1 criteria
OS（Overall Survival) | 2.5 years
  OS is the time interval from the date of randomization to death from any cause.
The incidence of AEs（adverse events) and SAEs（serious adverse events) | 2 years
  Frequency and severity of Adverse Events or Serious Adverse Events as defined by CTCAE version 5.0
ORR in subgroup of different TMB、PDL-1 and MSI status | 1.5 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria in subgroup of different TMB、PDL-1 and MSI status

OTHER OUTCOMES:
PK(pharmacokinetics) of envofolimab and BD0801 | 1.5 years
  Plasma concentrations of envofolimab an BD0801 will be measured.
Positive rate of ADA(anti-drug antibody) | 1.5 years
Duration of immunogenicity positive reaction | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhengguang Lv, Study Director — Jiangsu Simcere Pharmaceutical Co., Ltd.
Locations (24):
- China (24):
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Dezhou People'S Hospital, Dezhou
  - First Affiliated Hospital of Gannan Medical Universit, Ganzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Sun Yat-sen University affiliated with the Sixth Hospital, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Shaw Hospital Affiliated to Medical College of Zhejiang Universit, Hangzhou
  - Zhejiang Provincial People'S Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Chest Hospital, Hefei
  - Anhui Provincial Cancer Hospital, Hefei
  - The First Affliated Hospital Of Anhui Medical University, Hefei
  - Shandong Cancer Hospital, Jinan
  - Mianyang Central Hospital, Mianyang
  - Liaoning Cancer Hospital, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijia Zhuang
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Yantai Yuhuagnding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No